CLINICAL TRIAL: NCT04469166
Title: Effects of the Use of Tourniquet in Total Knee Arthroplasty on the Clinical and Functional Outcomes With 5 Years of Follow up: a Randomized Controlled Trial
Brief Title: Effects of the Use of Tourniquet in Total Knee Arthroplasty on the Clinical and Functional Outcomes With 5 Years of Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMU/Sherwan 10
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Use of Tourniquet in Total Knee Arthroplasty
Keywords: Tourniquet; Total knee arthroplasty; Clinical outcomes; Functional outcomes
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet (Active Comparator): Group of tourniquet
  Interventions: Procedure: tourniquet
- No tourniquet (Active Comparator): Group of no tourniquet
  Interventions: Procedure: No tourniquet

INTERVENTIONS:
Procedure: tourniquet — Use of tourniquet
  Arms: Tourniquet
Procedure: No tourniquet — No use of tourniquet
  Arms: No tourniquet

SUMMARY:
This study is randomized controlled trial with 5 years follow up and involved 101 patients divided in two groups; group A in which tourniquet was used in total knee arthroplasty while group B in which tourniquet was not used. All these patients were analyzed for the clinical and functional outcome measures.

DETAILED DESCRIPTION:
In this study, investigators have primary outcome measures and secondary outcome measures which were assessed in multiple periods to see the effects of using tourniquet in total knee arthroplasty on the clinical and functional outcomes with follow up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Grade 3 and 4 osteoarthritis
* age 55-80 years
* patients agree to participate in the study

Exclusion Criteria:

* Smoking
* Diabetes mellitus .Symptomatic spinal pathology with moderate to severe cervical or lumbosacral spinal stenosis.
* Hip pathology like osteoarthritis or fractures
* Neuromuscular disorders
* Blood dyscrasia or anticoagulant treatment .Body mass index equal to 30 or more.
* Previous knee surgery or knee infection
* Peripheral vascular disease
* Rheumatoid arthritis
* Hemoglobin less than 12 gram/deciliter

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Knee society score | This score was assessed at 5 years postoperatively
  Knee society score for functional outcome which will be low in poor function and high in best function
Knee injury and osteoarthritis outcome scores | This score was assessed at 5 years post-operatively
  Knee injury and osteoarthritis outcome score which will be low in poor function and high in better function
VAS for thigh pain | This score was assessed at 1st day post-operatively
  Visual analogue scale for thigh pain which will be high in more pain and low in less pain

SECONDARY OUTCOMES:
Post operative complications | These complications as bleeding, infection, Deep venous thrombosis and revision are assessed at postoperative period.
  The complications can occurred after surgery

IPD SHARING:
Plan to Share IPD: Undecided
Upon the publication of our study, I will decide to share my patients data